CLINICAL TRIAL: NCT00221117
Title: Neuroprosthesis for Improving Grasping Function in Spinal Cord Injured Patients
Brief Title: Benefits of Applying Neuroprosthesis to Improve Grasping and Reaching in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Christopher Reeve Paralysis Foundation (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Milos Popovic, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRI REB #02-032
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Occupational Therapy (COT) (Active Comparator): Conventional Occupational Therapy pertaining to hand function represents the current best practice activities against which the FET was compared. The COT included the following: (a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach; (b) task-specific, repetitive functional training; (c) strengthening and motor control training using resistance to available arm motion to increase strength; (d) stretching exercises; (e) electrical stimulation applied primarily for muscle strengthening (this was neither FES nor FET, but electro muscular stimulation); (f) practice of activities of daily living (ADLs) including self-care where the upper extremities were used as appropriate; and (g) caregiver training.
  Interventions: Other: Conventional Ocupational Therapy (COT)
- Neuroprosthesis-FES Therapy (Experimental): The FES Therapy began by designing stimulation protocols to generate power (circular grip and lateral pinch) and precision (opposition with 2 and 3 fingers) grasps on demand. The stimulation sequence (protocol) for power and precision grasps was developed for each patient individually using the Compex Motion electric stimulator. Compex Motion is a fully programmable transcutaneous (surface) stimulator that uses self-adhesive surface electrodes.
  Interventions: Device: Neuroprosthesis-FES Therapy

INTERVENTIONS:
Device: Neuroprosthesis-FES Therapy — The Compex Motion neuroprostesis, developed by Drs. R. Popovic and Thierry Keller,and company Compex SA, ia a flexible device designed to improve grasping function in both SCI and stroke patients.This multi-channel surface stimulation system for grasping provides both palmar and lateral grasp , and holds a number of advantages over the other existing neuroprostheses.
  Other Names: Neuroprosthesis
  Arms: Neuroprosthesis-FES Therapy
Other: Conventional Ocupational Therapy (COT) — Conventional occupational therapy pertaining to hand function represents control activities against which the FES therapy was assessed. The conventional occupational therapy included: a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach; b) task-specific, repetitive functional training; c) strengthening and motor control training using resistance to available arm motion to increase strength; d) stretching exercises; e) electrical stimulation applied primarily for muscle strengthening (this is not FES but TENS application); f) activities of daily living including self-care where the upper limb was used as an assist if appropriate; and g) caregiver training.
  Other Names: Conventional Occupational Therapy (COT)
  Arms: Conventional Occupational Therapy (COT)

SUMMARY:
Functional electrical stimulation is a process that uses low intensity electrical pulses generated by an electric stimulator to create muscle contractions. By contracting muscles in a specific sequence, one can generate various body functions such as grasping, walking, and standing.The study is designed to evaluate the effectiveness and long term benefits of applying functional electrical simulation during early rehabilitation to improve grasping function in persons who have suffered a spinal cord injury. By using functional electrical stimulation,these patients could potentially improve their grasping function.

DETAILED DESCRIPTION:
The main objective of this study is to determine the effectiveness of a new treatment regime that uses a neuroprosthesis for the improvement and recovery of grasping functions in persons with spinal cord injuries (SCI). This treatment has been shown to be useful for stroke patients with hemiplegic arm in the recovery of reaching and grasping 1, and our preliminary work indicates that this may also be the case with SCI patients 3. Further, aside from the potential of promoting voluntary grasp in SCI patients, this novel therapeutic approach may also impact the way service is currently delivered in SCI rehabilitation settings.

A neuroprosthesis for grasping is a device that can improve or restore the grasping, holding, and releasing functions in persons with SCI 2, 3. The neuroprosthesis applies functional electrical stimulation (FES) to artificially generate a muscle contraction by applying short current pulses to motor nerves innervating muscles. FES can be applied to individuals with incomplete SCI to help them restore functions such as walking and grasping by contracting groups of paralyzed muscles in an orchestrated manner 4. FES was originally envisioned as an intervention that was 'permanent' in nature. In other words, an individual had to wear/use an FES orthotic device at all times if s/he wanted to generate the function that was impaired by SCI 4. Our application of the neuroprosthesis for grasping in this proposal presents a departure from this standard and established approach of FES application. Rather than having people be dependent on the neuroprosthesis to perform their activities of daily living (ADL), we plan to use the neuroprosthesis for grasping as a short-term intervention that will help SCI individuals recover voluntary grasping function. Hence, we believe that those participants who undergo our FES therapy with the neuroprosthesis should be able to perform grasping functions without its use once the treatment program is completed.

Recent innovative advances in FES applications, spearheaded by our team, clearly indicate that the short-term, therapeutic intervention of the neuroprosthesis for grasping can enhance voluntary function in individuals with SCI 3, 5, 6. These studies also suggest that this novel method of applying FES to augment functional improvement has the potential to improve overall physical and psychological well being of persons with incomplete SCI. Since 1999, the Co-PI of this application, Dr. Milos Popovic and Dejan Popovic's team from the University of Belgrade have reported anecdotal evidence that some C5 to C7 SCI individuals who were unable to voluntarily grasp, were later able to do so after intensive training with a neuroprosthesis for grasping 2, 7, 8, 9. They observed that approximately 20 to 25% of the individuals who trained with the FES systems were able to grasp without the assistance of the neuroprosthesis once the systems were removed. Although this evidence has been presented in several peer-reviewed publications, there have been no comprehensive studies to date that have investigated the long-term effects of FES treatment on recovery of the voluntary grasping function in persons with SCI. Consequently, this study seeks to 1) investigate whether a series of orchestrated FES therapies can be applied to re-train/improve voluntary grasping function in acute SCI individuals, and; 2) to determine whether this therapy will yield better results than conventional occupational therapy. Specifically, we will recruit participants who have C5 to C7 incomplete SCI. These individuals typically can generate weak wrist extension but can neither flex, extend, abduct or adduct the fingers, nor flex, extend, abduct or adduct the thumb. Our therapy will be used to help these individuals recover some or all of these functions.

ELIGIBILITY:
Inclusion Criteria:

* traumatic spinal cord lesion between C4 and C7(incomplete)
* participants will be recruited during the first six months post-SCI.

Exclusion Criteria:

* uncontrolled hypertension
* susceptibility to autonomic dysreflexia
* pressure ulcer
* cardiac pacemakers
* skin rush

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milos Popovic, Ph.D, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared , mean results of the study have been published in the peer reviewed paper.

REFERENCES:
- [Background] Popovic MR, Curt A, Keller T, Dietz V. Functional electrical stimulation for grasping and walking: indications and limitations. Spinal Cord. 2001 Aug;39(8):403-12. doi: 10.1038/sj.sc.3101191. PMID 11512070
- [Derived] Kapadia NM, Bagher S, Popovic MR. Influence of different rehabilitation therapy models on patient outcomes: hand function therapy in individuals with incomplete SCI. J Spinal Cord Med. 2014 Nov;37(6):734-43. doi: 10.1179/2045772314Y.0000000203. Epub 2014 Jun 26. PMID 24968955
- See also: Rehabilitation Engineering Laboratory — http://www.toronto-fes.ca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized using 2 sets of sealed envelopes. Each unmarked envelope contained a single sheet of paper with a printed number in the range of 1 to 40. A second set of envelopes was marked with numbers from 1 to 40 and contained a single sheet specifying the group allocation.
Pre-assignment Details: If participant did not meet inclusion criteria they would be excluded
Groups:
- Conventional Occupational Therapy-Control Group: Conventional occupational therapy pertaining to hand function represents control activities against which the FES therapy was assessed. The conventional occupational therapy included: a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach; b) task-specific, repetitive functional training; c) strengthening and motor control training using resistance to available arm motion to increase strength; d) stretching exercises; e) electrical stimulation applied primarily for muscle strengthening (this is not FES but TENS application); f) activities of daily living including self-care where the upper limb was used as an assist if appropriate; and g) caregiver training.
- Fes Therapy-Treatment Group: The FET began by designing stimulation protocols to generate power (circular grip and lateral pinch) and precision (opposition with 2 and 3 fingers) grasps on demand. The stimulation sequence (protocol) for power and precision grasps was developed for each patient individually using the Compex Motion electric stimulator. Compex Motion is a fully programmable transcutaneous (surface) stimulator that uses self-adhesive surface electrodes.
Period: Overall Study
Arm/Group | Conventional Occupational Therapy-Control Group | Fes Therapy-Treatment Group
Started | 12 | 9 (One participant dropped out of the study after signing consent but prior to baseline assessments.)
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Occupational Therapy-Control Group | Fes Therapy-Treatment Group | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.75 (4.72) | 43.2 (5.45) | 43.975 (5.085)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Functional Independence Measure (FIM)
Description: Functional Independent Measure was employed to measure the degree of disability for daily self care. It capture data on self-care, sphincter management, transfers,locomotion,communication,and social cognition.The scale is divided according to no helper category (level 6 and 7) where no other person is required to help with the activity and a hel;per category(level 1 through 5)where the patient needs minimal to total assistance from another person to accomplish the activity Score range from 18-126. Higher values represent a better outcome.
Time Frame: 35 min
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FES Therapy; Conventional Occupational Therapy: The Functional Independence Measure (FIM)15 was employed to measure the degree of disability for daily self-care.
Arm/Group | FES Therapy | Conventional Occupational Therapy
Number analyzed (Participants) | 9 | 12
units on a scale | 20.1 (9.87) | 10 (9.065)
Statistical Analysis 1: Comparison: FES Therapy vs Conventional Occupational Therapy; Test type: Other; p = .015, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Rehabilitation Engineering Laboratory Hand Function Test(REL Test)
Description: The Toronto Rehabilitation Institute Hand Function Test (TRI-HFT) evaluates gross motor function of unilateral grasp (also referred to as the Rehabilitation Engineering Laboratory Hand Function Test). Hand functions that are assessed with TRI-HFT include the following: lateral or pulp pinch and palmar grasp.Score range from 0-70. Higher values represent a better outcome.
Time Frame: 45 min
Population: The subject's impairment and demographic characteristics were analyzed using descriptive statistics for parametric and nonparametric data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FES Group | Conventional Occupational Therapy
Number analyzed (Participants) | 9 | 12
units on a scale | 16.7 (14.80) | 11.3 (9.52)
Statistical Analysis 1: Comparison: FES Group; The subject's impairment and demographic characteristics were analyzed using descriptive statistics for parametric and nonparametric data. The baseline outcome data of the intervention and control groups were compared using Fisher exact test (for categorical variables) and Mann-Whitney U test (for continuous variables). Comparisons between the intervention and control groups were carried out using linear regression analysis adjusted for the baseline degree of disability (baseline AIS); Test type: Superiority or Other; p = 0.05, Regression, Linear

3. Secondary Outcome: Spinal Cord Independence Measure (SCIM).
Description: Score range from 0-100. Higher score represent a better outcome.
Time Frame: 30 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FES Therapy | Conventional Occupational Therapy
Number analyzed (Participants) | 9 | 12
units on a scale | 10.1 (3.8) | 3.1 (2.4)

ADVERSE EVENTS:
Groups:
- Control Group: Conventional Occupational Therapy
Arm/Group | Control Group | Fes Therapy-Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

LIMITATIONS AND CAVEATS:
A limitation of this study is that despite considerable effort we failed to attract the subjects to take part in a 6-month follow- up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No